CLINICAL TRIAL: NCT00488241
Title: A Multicenter, Open Uncontrolled Clinical Study to Examine the Efficacy and Safety of Zarzenda in the Management of Hand Eczema
Brief Title: Multicenter Clinical Study to Examine the Efficacy and Safety of Zarzenda in Patients With Hand Eczema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1401663; NCT01646658 (obsolete NCT alias)
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hand Eczema
Keywords: Eczema; Medical device
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Topically applied daily for 2 weeks
  Interventions: Device: Zarzenda

INTERVENTIONS:
Device: Zarzenda — Topically applied daily for 2 weeks

SUMMARY:
To show efficacy of Zarzenda in the treatment of hand eczema

DETAILED DESCRIPTION:
The objective of the study is to demonstrate efficacy and safety of Zarzenda (a medical device) in the management of hand eczema.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hand eczema for at least 3 months
* At least 4 weeks have passed since use of systemic treatment for eczema
* At least 4 weeks have passed since any vaccination
* At least 1 week has passed since last topic treatment on hands with corticosteroids
* Agree to use adequate contraceptive method if of childbearing potential
* Willingness to avoid excessive exposure to sunlight and avoid skin irritants

Exclusion Criteria:

* Pregnancy, breast feeding
* Severe excoriations on the hands
* Need for systemic treatment for atopic dermatitis
* Known sensitivity to Zarzenda and/or to extract of nut butyrospermum parkii (shea)
* Known immune deficiency
* Concomitant infection on hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Hand eczema severity index (HECSI)at the end of study | End of study compared to baseline

SECONDARY OUTCOMES:
Investigator's Global Assessment | End of study compared to baseline
Patients assessment of itch | End of study compared to baseline
Hand surface area | End of study compared to baseline
Clinical signs of hand eczema | End of study compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Intendis GmbH, Berlin, Germany